CLINICAL TRIAL: NCT01036412
Title: Chlorhexidine Gel Therapy for Cariogenic Oral Microflora in Irradiated Head and Neck Cancer Patients
Brief Title: Chlorhexidine Gel Therapy for Cariogenic Oral Microflora
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-0456
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2012-08

CONDITIONS: Head and Neck Cancer
Keywords: Chlorhexidine; Chlorhexidine Gel Therapy; 1% chlorhexidine gluconate gel; Cariogenic Oral Microflora; Irradiated Head and Neck Cancer Patients; caries-forming organisms; Radiation treatment; Mouth Cancer; Throat Cancer; Tooth decay
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Dental Caries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chlorhexidine Gel Therapy (Experimental): Following 2 x 5-minute applications of 2.5 ml in clinic, 2 x 5.0 ml syringes of 1% chlorhexidine gluconate gel, self-administered for a 5-minute application Week 2 & Week 4
  Interventions: Drug: 1% Chlorhexidine Gluconate Gel; Behavioral: Surveys

INTERVENTIONS:
Drug: 1% Chlorhexidine Gluconate Gel — Following two 2.5 ml 5-minute applications performed in clinic on Day 1, 2 x 5.0 ml syringes of chlorhexidine gel self-administered for one 5-minute application using the custom-made carriers carriers on week 2 (12-14 days from baseline visit study drug administration) and week 4 (12-14 days from Week 2 study drug administration).
  Other Names: Chlorhexidine Gel
Behavioral: Surveys — M. D. Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) questionnaire, in addition to a 2nd subjective, study-specific questionnaire administered during visit taking about 5 minutes to complete each assessment.
  Other Names: Questionnaire

SUMMARY:
The goal of this clinical research study is to find out if 1% chlorhexidine gluconate gel will decrease the amount of bacteria that causes tooth decay. Whether the gel is acceptable to patients will also be studied.

DETAILED DESCRIPTION:
1% chlorhexidine gluconate gel is an alcohol-free, raspberry-flavored brush-on gel. It is designed to decrease the amount of bacteria found in your mouth that can cause tooth decay.

Within a month, if you are found to be eligible to take part in this study, researchers will use custom dental trays designed for you, in order to deliver the chlorhexidine gel. During your next visit to the dental clinic, researchers will place these custom dental trays and the gel in your mouth for about 5 minutes. Over the next 30 minutes, the gel will be applied one more time. The dentist will also chart your decayed, missing, and filled teeth in a dentist chart during this visit. The dentist will also check the soft tissues of your mouth. You will have an office visit the next day (Day 2) to see if you had any side effects to the chlorhexidine gel.

These trays will be coated with the gel every 2 weeks, for a 12-week period. You will hold the trays with the gel in your mouth for at least 5 minutes, usually at night or in the morning. You should not eat or drink during these 5 minutes in order to increase the effectiveness of the gel on your teeth. You will apply the gel at home, for one 5-minute application, on Weeks 2, 4, 8 and 10. You will be given a diary to list each time that you use the gel at home, and to list if you experience any side effects. You will have office visits on Weeks 6 and 12. The dentist will floss between all of your teeth during these office visits. You will also use the gel, for two 5-minute applications, during these office visits. You will also need to bring the completed diary to each office visit.

When you return for the office visit, a dentist or dental hygienist will then collect a sample of your dental plaque (a film of mucous and bacteria found on your teeth's surface) by scraping plaque from the surface of your teeth and flossing between your teeth, and then placing the plaque in a small test tube to check for bacteria. The dentist will not scrape below the gums. These plaque samples will be collected on Weeks 6 and 12 at the dental clinic.

Once the gel application period is over, you will need to return to the dental clinic for plaque sample scrapings at Weeks 16 and 20 so that researchers can check to see if the bacteria is growing again.

You will also complete two questionnaires during your baseline, Week 6, and Week 12 visits to describe your experience with the use of the gel and your side effects from radiation treatment.

Once your last plaque sample scraping has been collected on Week 20, your participation in this study will be complete. The dentist or dental hygienist will floss between all of your teeth and your decayed, missing, and filled teeth will be charted in a dentist chart during the Week 20 office visit. You will be taken off study if intolerable side effects occur.

This is an investigational study. 1% chlorhexidine gluconate is not FDA approved or commercially available. It has been authorized for use in research only. About 50 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

1. Patients who have undergone radiation treatment to the head and neck at U.T. M. D. Anderson Cancer Center for oral cavity or oropharyngeal cancer (base of tongue and tonsil) and have recent documented caries, within 8 weeks, on routine oral examination.
2. Patients with >/= 10 teeth.
3. Patients with >/= 100,000 CFU/ ml S. mutans in the baseline microbiological sample (i.e., supragingival curette sampling).

Exclusion Criteria:

1. Patients using antibiotics in the past 4 weeks. (Note: A subject may have antibiotics administered during the study evaluation period, for unforeseen medical reasons. The patients will not be removed from the study and the plaque samples will be evaluated for descriptive assessment with the concomitant medication(s) recorded to determine if changes between the subject's samples were globally outside the range of changes for the population as a whole.)
2. Patients using chlorhexidine gluconate or antimicrobial rinses in past 2 weeks.
3. Patients under the age of 18.
4. Patients unable to return to dental clinic over the 20-week study period.
5. Patients with a known allergy to Chlorhexidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Microbiology Assessments (Evaluation of colony forming units of Streptococcus mutans, Lactobacilli spp. and Actinomyces naeslundii and Actinomyces viscous) | 20 weeks
  At baseline, after initial drug administration, and on weeks 6 and 12 of drug administration; and weeks 16 and 20 after cessation of drug application.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda F. Jacob, MS, BS, DDS, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org